CLINICAL TRIAL: NCT00316017
Title: Phase 3 Study of Hypertonic Resuscitation Following Traumatic Injury With Hypovolemic Shock
Brief Title: Hypertonic Resuscitation Following Traumatic Injury
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility & potential safety concern (increased early mortality in the HS/HSD arms for those with no PRBC in 1st 24 hr, post-randomization subgp)
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); The Institute of Circulatory and Respiratory Health (ICRH) (Unknown); Defence Research and Development Canada (Industry)
Responsible Party: Gerald van Belle, PhD/Prinicipal Investigator, Resuscitation Outcomes Consortium Data Coordinating Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28226-A - IND 12506; 5U01HL077863-05 (NIH); IND #12506 (shock cohort) (Other: FDA)
Record Dates: First submitted 2006-04-17; First posted 2006-04-19 (Estimated); Results first posted 2010-11-11 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Shock, Traumatic
Keywords: Trauma; Shock
MeSH Terms: conditions — Shock, Traumatic; Wounds and Injuries; Shock | interventions — Saline Solution, Hypertonic; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 7.5% hypertonic saline/6% Dextran-70 (HSD)
  Interventions: Drug: 7.5% hypertonic saline/6% Dextran-70 (HSD)
- 2 (Experimental): 7.5% hypertonic saline (HS)
  Interventions: Drug: 7.5% hypertonic saline (HS)
- 3 (Placebo Comparator): 0.9% normal saline
  Interventions: Drug: 0.9% normal saline

INTERVENTIONS:
Drug: 7.5% hypertonic saline/6% Dextran-70 (HSD) — 250 cc dose given as a one-time intravenous (IV) bolus in the pre-hospital setting.
  Other Names: RescueFlo
  Arms: 1
Drug: 7.5% hypertonic saline (HS) — 250 cc dose given as a one-time IV bolus in the pre-hospital setting.
  Arms: 2
Drug: 0.9% normal saline — 250 cc dose given as a one-time IV bolus in the pre-hospital setting.
  Arms: 3

SUMMARY:
The purpose of this study is to determine if hypertonic saline with and without dextran can improve overall survival in victims of trauma with shock.

Injury and lost blood from trauma can cause your body to be in shock (low blood pressure related to blood loss). This decreased blood flow can lead to organ damage. In order to restore the blood pressure and blood flow, the medics give fluids into the patients' veins as soon as possible. This is called "resuscitation." The resuscitation fluid most commonly used is "isotonic" or one that is the same concentration as the blood. The investigators are trying to determine if infusing a "hypertonic" fluid (or one more concentrated than the blood) can increase the blood pressure and restore blood flow more efficiently. The hypertonic fluids the investigators are using are called hypertonic saline with dextran (HSD) and hypertonic saline (no dextran). Hypertonic saline is a salt solution that is slightly more concentrated than your blood. Dextran is a sugar solution.

DETAILED DESCRIPTION:
Specific Aim: To determine if prehospital administration of 7.5% hypertonic saline /6% Dextran-70 (HSD) OR 7.5% hypertonic saline alone (HS), compared to current standard therapy with normal saline (NS), as an initial resuscitation fluid, affects survival following traumatic injury with hypovolemic shock.

Trauma is the leading cause of death among North Americans between the ages of 1 and 44 years. The majority of these deaths result from hypovolemic shock or severe brain injury. Patients in hypovolemic shock develop a state of systemic tissue ischemia then a subsequent reperfusion injury at the time of fluid resuscitation. Conventional resuscitation involves the IV administration of a large volume of isotonic or slightly hypotonic (lactated ringers, LR) solutions beginning in the prehospital setting. Although not conclusive, prior studies have suggested that alternative resuscitation with hypertonic saline (7.5%) solutions may reduce morbidity or mortality in these patients. Furthermore, hypertonic fluids may have specific advantages in the brain-injured patient, as they may aid in the rapid restoration of cerebral perfusion and prevent extravascular fluid sequestration, thereby limiting secondary brain injury. In addition, recent studies have demonstrated that hypertonicity significantly alters the activation of inflammatory cells, an effect that may reduce subsequent organ injury from ischemia-reperfusion and decrease nosocomial infection. The majority of previous clinical trials have focused on the use of HSD. The potential for 7.5% saline alone (HS) to have similar effects has not been well studied. Removal of the dextran component may enhance the anti-inflammatory effects of this solution, which could improve secondary outcomes such as acute respiratory distress syndrome (ARDS), multiple organ failure syndrome (MOFS) and rates of nosocomial infections.

This study is a randomized, double-blind, three-arm placebo controlled trial designed to evaluate the clinical outcome of trauma patients with hypovolemic shock, as manifested by prehospital hypotension. Patients will be randomized to a single 250cc IV dose of 7.5% saline in 6% Dextran-70 (HSD), 7.5% saline (HS) or normal saline as the initial fluid for prehospital resuscitation. No additional interventions will occur once the patient is admitted to the hospital. In hospital data collection will last up to 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Blunt or penetrating trauma
* Prehospital Systolic Blood Pressure (SBP) <= 70;OR
* Prehospital SBP 71-90 AND Hear Rate (HR) ≥108
* 15 years of age or older, or 50kg or more if age unknown

Exclusion Criteria:

* Known or suspected pregnancy
* Age younger than 15 or less than 50kg if age unknown
* Ongoing prehospital cardiopulmonary resuscitation (CPR)
* Administration of more than 2000cc crystalloid or any colloid or blood products
* Severe hypothermia (suspected Temperature less than 28 degrees celsius)
* Drowning or asphyxia due to hanging
* Burns Total Body Surface Area (TBSA) more than 20%
* Isolated penetrating injury to the head
* Inability to obtain prehospital intravenous access
* Time of call received at dispatch to study intervention greater than four hours
* Known prisoners

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 895 (Actual)
Dates: Start 2006-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron L Weisfeldt, MD, Study Chair — Resuscitation Outcomes Consortium
Locations (10):
- United States (8):
  - Alabama Resuscitaion Center, University of Alabama, Birmingham, Alabama
  - UCSD-San Diego Resuscitation Research Center, San Diego, California
  - Iowa Resuscitation Network, University of Iowa Carver College of Medicine, Iowa City, Iowa
  - Portland Resuscitation Outcomes Consortium, Oregon Health & Sciences University, Portland, Oregon
  - The Pittsburgh Resuscitation Network, University of Pittsburgh, Pittsburgh, Pennsylvania
  - Dallas Center for Resuscitation Research, University of Texas Southwestern Medical Center, Dallas, Texas
  - Seattle-King County Center For Resuscitation Research, University of Washington, Seattle, Washington
  - Milwaukee Resuscitation Network, Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - University of Ottawa/University of British Columbia Collaborative RCC, Ottawa Health Research Institute, Ottawa, Ontario
  - Toronto Regional Resuscitation Research Out-of-Hospital Network, University of Toronto, Toronto, Ontario

REFERENCES:
- [Result] Bulger EM, May S, Kerby JD, Emerson S, Stiell IG, Schreiber MA, Brasel KJ, Tisherman SA, Coimbra R, Rizoli S, Minei JP, Hata JS, Sopko G, Evans DC, Hoyt DB; ROC investigators. Out-of-hospital hypertonic resuscitation after traumatic hypovolemic shock: a randomized, placebo controlled trial. Ann Surg. 2011 Mar;253(3):431-41. doi: 10.1097/SLA.0b013e3181fcdb22. PMID 21178763
- [Derived] Tisherman SA, Schmicker RH, Brasel KJ, Bulger EM, Kerby JD, Minei JP, Powell JL, Reiff DA, Rizoli SB, Schreiber MA. Detailed description of all deaths in both the shock and traumatic brain injury hypertonic saline trials of the Resuscitation Outcomes Consortium. Ann Surg. 2015 Mar;261(3):586-90. doi: 10.1097/SLA.0000000000000837. PMID 25072443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled by Emergency Medicine Services (EMS) personnel in the pre-hospital setting based on pre-defined inclusion/exclusion criteria. The first subject was enrolled on May 9, 2006 and the last subject was enrolled on August 25, 2008.
Pre-assignment Details: 895 subjects were randomized. 852 subjects completed the study. Randomization was performed when the outer study fluid bag wrapper was removed in the presence of a patient. To ensure there was no bias, a secondary intention to treat analysis was also performed which included all randomized patients even if the fluid was not administered.
Groups:
- 7.5% Hypertonic Saline/6% Dextran-70 (HSD): 7.5% hypertonic saline/6% Dextran-70 (HSD) 250 ml
- 7.5% Hypertonic Saline (HS): 7.5% hypertonic saline (HS) 250ml dose
- 0.9% Normal Saline: 0.9% normal saline 250 ml dose as placebo
Period: Overall Study
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Started | 231 (11 of 11 not completed due to "Bag Opened Not Given" (BONG)) | 269 (12 of 13 not completed due to BONG; 1 not completed was a prisoner who was excluded) | 395 (19 of 19 not complete due to BONG)
Completed | 220 | 256 | 376
Not Completed | 11 | 13 | 19
Not completed — Protocol Violation | 11 | 13 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline | Total
Number analyzed (Participants) | 220 | 256 | 376 | 852
Age Categorical [Number; unit: participants] — The HSD group included one subject with no age data available.
  participants
    <=18 years | 13 | 13 | 23 | 49
    Between 18 and 65 years | 188 | 225 | 332 | 745
    >=65 years | 18 | 18 | 21 | 57
Age Continuous [Mean (Standard Deviation); unit: years] — The HSD group included one subject with no age data available.
  years | 37.7 (17.3) | 36.8 (16.1) | 36.2 (16.4) | 36.7 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Description only includes those subjects who received the study fluid.
  Participants
    Female | 50 | 51 | 85 | 186
    Male | 170 | 205 | 291 | 666
Region of Enrollment [Number; unit: participants]
  United States | 177 | 212 | 283 | 672
  Canada | 43 | 44 | 93 | 180

OUTCOME MEASURES:

1. Primary Outcome: 28 Day Survival
Description: The day of episode is counted as "Day 0". So for measures using a 28 day period, the maximum value is 29 (i.e. days 0 through 28).
Time Frame: 28 days from time of Emergency Department (ED) arrival
Population: Per protocol, analysis was done on only those subjects who received the study fluid per randomization; this was defined as that the study fluid had been connected to the patient's IV.
Measure: Number; unit: participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 220 | 256 | 376
participants | 164 | 187 | 279
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in the percent of patients who survived to day 28 day between the three groups; Test type: Superiority or Other; p = 0.91, test for proportions — The Statistical Analysis applies to the 7.5% hypertonic saline/6% Dextran-70 (HSD),7.5% hypertonic saline (HS), and 0.9% normal saline groups

2. Secondary Outcome: Adult Respiratory Distress Syndrome(ARDS)-Free Survival Through Day 28
Description: Absence of diagnosis of Adult Respiratory Distress Syndrome and alive through day 28
Time Frame: 28 days from time of ED arrival
Measure: Number; unit: participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 220 | 256 | 376
participants | 147 | 170 | 246
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in ARDS-free survival through day 28 between the three groups; Test type: Superiority or Other; p = 0.94, test for proportions — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Worst Multiple Organ Dysfunction Score (MODS) Mean Through Day 28
Description: Multiple Organ Dysfunction Score is described as:
  Six organ systems were chosen, and a score of 0-4 allotted for each organ according to function (0 being normal function through to 4 for most severe dysfunction) with a maximum score of 24. The worst score based on available data (missing values were assumed normal) in each 24-hour period is taken for calculation of the aggregate score.
Time Frame: 28 days from time of ED arrival
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 220 | 256 | 376
Scores on a scale | 8.7 (9.8) | 9.3 (9.6) | 8.8 (9.7)
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in average Worst Multiple Organ Dysfunction Scores (MODS) through day 28 between the three groups; Test type: Superiority or Other; p = 0.73, ANOVA — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Presence of Nosocomial Infection Through Day 28
Description: Includes one or more nosocomial infections from the following list: pneumonia, blood stream infection, urinary tract infection and wound infection
Time Frame: Within 28 days of injury, while hospitalized
Measure: Number; unit: participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 220 | 256 | 376
participants | 52 | 63 | 89
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in the percent of patients with the Presence of Nosocomial Infection through day 28 between the three groups; Test type: Superiority or Other; p = 0.8, test for proportions — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Packed Red Blood Cells (PRBC) First 24 Hours
Description: The numbers of units of packed red blood cells transfused in the first 24 hours
Time Frame: First 24 hours from the time of 911 call
Measure: Mean (Standard Deviation); unit: units of packed red blood cells
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 220 | 256 | 376
units of packed red blood cells | 4.81 (8.12) | 4.61 (7.46) | 5.15 (8.29)
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in the average number of PRBC units given within the first 24 hours between the three groups; Test type: Superiority or Other; p = 0.69, ANOVA — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: Total Fluids First 24 Hours
Description: The total amount of IV fluids given in the pre-hospital setting and the hospital setting in the first 24 hours following the time of 911 call
Time Frame: First 24 hours from the time of of 911 call
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 220 | 256 | 376
Liters | 11.4 (9.6) | 11.6 (10.4) | 12.3 (12.1)
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in the average amount of Total fluids given within the first 24 hours between the three groups; Test type: Superiority or Other; p = 0.57, ANOVA — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Ventilator-free Days Through Day 28
Description: The number of days beginning with the day of 911 call counted as "Day O" through day 28 that the patient did not require mechanical ventilation
Time Frame: Duration of hospital stay through day 28
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 220 | 256 | 376
days | 18 (12.3) | 17 (12.2) | 17.5 (12.4)
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in the average number of Ventilator-free days through day 28 between the three groups; Test type: Superiority or Other; p = 0.66, ANOVA — [p-value comment as in outcome 1, analysis 1]

8. Secondary Outcome: Days Alive Out of the Intensive Care Unit (ICU) Through Day 28
Description: The number of days the patient is alive and not being cared for in the intensive care unit
Time Frame: First 28 days from the time of 911 call
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 220 | 256 | 376
days | 16.4 (12.3) | 15.7 (12.0) | 16 (12.2)
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in the average number of Days alive out of the ICU through day 28 between the three groups; Test type: Superiority or Other; p = 0.82, ANOVA — [p-value comment as in outcome 1, analysis 1]

9. Secondary Outcome: Days Alive Out of the Hospital Through Day 28
Description: The number of days the patient is alive and no longer an inpatient in the hospital through day 28
Time Frame: First 28 days from the time of 911 call
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 220 | 256 | 376
days | 10.3 (10.7) | 10.3 (10.8) | 10.1 (10.6)
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in the average number of Days alive out of the hospital through day 28 between the three groups; Test type: Superiority or Other; p = 0.98, ANOVA — [p-value comment as in outcome 1, analysis 1]

10. Secondary Outcome: Survival at Hospital Discharge
Description: Alive at the time of discharge from the Level One or Two trauma hospital. This did not include disposition from rehabilitation facilities.
Time Frame: Duration of hospital stay through to discharge
Measure: Number; unit: participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 220 | 256 | 376
participants | 163 (26.3) | 185 (28.3) | 278 (27.5)
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in the percent of patients who survived to hospital discharge between the three groups; Test type: Superiority or Other; p = 0.85, test for proportions — [p-value comment as in outcome 1, analysis 1]

11. Secondary Outcome: Zero Units PRBC in First 24 Hours
Description: This is the total number of subjects who received no blood products in the first 24 hours from the time of the 911 call.
Time Frame: From the time dispatch received the 911 call to the end of the first 24 hours
Measure: Number; unit: participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 220 | 256 | 376
participants | 91 | 104 | 139
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in the percent of patients who received zero units of PRBC in the first 24 hours between the three groups; Test type: Superiority or Other; p = 0.48, test for proportions — [p-value comment as in outcome 1, analysis 1]

12. Secondary Outcome: Zero Units PRBC and Died in Field or Emergency Department (ED)
Description: This is the total number of subjects who died in the field or the ED from the set of subjects who received no blood products.
Time Frame: From the time dispatch received 911 call to the time of death in the field or ED
Measure: Number; unit: participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 91 | 104 | 139
participants | 14 | 23 | 13
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in the percent of patients who died in field or ED between the three groups among the patients who received zero units of PRBC; Test type: Superiority or Other; p < 0.01, test for proportions — [p-value comment as in outcome 1, analysis 1]

13. Secondary Outcome: Zero Units PRBC and Died Within 6 Hours of Admission to the Hospital
Description: This is the total number of subjects who died within the first 6 hours from the time of admission to the hospital among the patients who received no blood products.
Time Frame: The first 6 hours from the time of admission to the hospital
Measure: Number; unit: participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 91 | 104 | 139
participants | 15 | 23 | 14
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in percent of patients who died within 6 hours of admission to the hospital between the three groups among patients who received zero units of PRBC; Test type: Superiority or Other; p < 0.02, test for proportions — [p-value comment as in outcome 1, analysis 1]

14. Secondary Outcome: Zero Units PRBC and Died Within 28 Days From the Time of the 911 Call
Description: This is the total number of subjects who died within 28 days from the time of the 911 call among the patients who received no units of PRBC.
Time Frame: From the time dispatch received the 911 call to 28 days
Measure: Number; unit: participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 91 | 104 | 139
participants | 22 | 31 | 18
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in the percent of patients who died within 28 days from the time of the 911 call between the three groups among the patients who received zero units of PRBC; Test type: Superiority or Other; p < 0.01, test for proportions — [p-value comment as in outcome 1, analysis 1]

15. Secondary Outcome: 1-9 Units PRBC in First 24 Hours
Description: This is the total number of subjects who received 1 to 9 units of packed red blood cells (PRBC) in the first 24 hours from the time of the 911 call.
Time Frame: From the time dispatch received the 911 call to the end of the first 24 hours
Measure: Number; unit: participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 220 | 256 | 376
participants | 92 | 111 | 175
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in the percent of patients who received 1-9 units PRBC in the first 24 hours between the three groups; Test type: Superiority or Other; p = 0.51, test for proportions — [p-value comment as in outcome 1, analysis 1]

16. Secondary Outcome: 1-9 Units PRBC and Died in Field or ED
Description: This is the total number of subjects who received 1 to 9 units of packed red blood cells (PRBC) among the patients who died in the field or the ED.
Time Frame: From the time dispatch received 911 call to the time of death in the field or ED
Measure: Number; unit: participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 92 | 111 | 175
participants | 11 | 10 | 14
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in the percent of patients who died in Field or ED between the three groups among the patients who received 1-9 units of PRBC; Test type: Superiority or Other; p = 0.73, test for proportions — [p-value comment as in outcome 1, analysis 1]

17. Secondary Outcome: 1-9 Units PRBC and Died Within 6 Hours of Admission to the Hospital
Description: This is the total number of subjects who died within the first 6 hours from the time of admission to the hospital among the patients who received 1 to 9 units of packed red blood cells (PRBC).
Time Frame: The first 6 hours from the time of admission to the hospital
Measure: Number; unit: participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 92 | 111 | 175
participants | 12 | 17 | 25
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in the percent of patients who died within 6 hours of admission to the hospital between the three groups among the patients who received 1-9 units of PRBC; Test type: Superiority or Other; p = 0.83, test for proportions — [p-value comment as in outcome 1, analysis 1]

18. Secondary Outcome: 1-9 Units PRBC and Died Within 28 Days From the Time of the 911 Call
Description: This is the total number of subjects who died within 28 days from the time of the 911 call among the patients who received 1 to 9 units of packed red blood cells (PRBC).
Time Frame: From the time dispatch received the 911 call to 28 days
Measure: Number; unit: participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 92 | 111 | 175
participants | 19 | 24 | 46
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in the percent of patients who died within 28 days from the time of the 911 call between the three groups among the patients who received 1-9 units of PRBC; Test type: Superiority or Other; p = 0.31, test for proportions — [p-value comment as in outcome 1, analysis 1]

19. Secondary Outcome: Greater Than 10 Units PRBC in First 24 Hours
Description: This is the total number of subjects who received greater than 10 units of packed red blood cells (PRBC) in the first 24 hours from the time of the 911 call.
Time Frame: From the time dispatch received the 911 call to the end of the first 24 hours
Measure: Number; unit: participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 220 | 256 | 376
participants | 36 | 40 | 61
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in the percent of patients who received greater than 10 units of PRBC in first 24 hours between the three groups; Test type: Superiority or Other; p = 0.97, test for proportions — [p-value comment as in outcome 1, analysis 1]

20. Secondary Outcome: Greater Than 10 Units PRBC and Died in Field or ED
Description: This is the total number of subjects who died in the field or the ED among the patients who received greater than 10 units of packed red blood cells (PRBC).
Time Frame: From the time dispatch received 911 call to the time of death in the field or ED
Measure: Number; unit: participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 36 | 40 | 61
participants | 0 | 0 | 3

21. Secondary Outcome: Greater Than 10 Units PRBC and Died Within 6 Hours of Admission to the Hospital
Description: This is the total number of subjects who died within the first 6 hours from the time of admission to the hospital among the patients who received greater than 10 units of packed red blood cells (PRBC).
Time Frame: The first 6 hours from the time of admission to the hospital
Measure: Number; unit: participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 36 | 40 | 61
participants | 9 | 9 | 22
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in the percent of patients who died within 6 hours of admission to the hospital between the three groups among the patients who received greater than 10 units of PRBC; Test type: Superiority or Other; p = 0.35, test for proportions — [p-value comment as in outcome 1, analysis 1]

22. Secondary Outcome: Greater Than 10 Units PRBC and Died Within 28 Days From the Time of the 911 Call
Description: This is the total number of subjects who died within 28 days from the time of the 911 call among the patients who received greater than 10 units of packed red blood cells (PRBC).
Time Frame: From the time dispatch received the 911 call to 28 days
Measure: Number; unit: participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Number analyzed (Participants) | 36 | 40 | 61
participants | 15 | 14 | 32
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran-70 (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline; The null hypothesis is that there are no differences in the percent of patients who died within 28 days from the time of the 911 call between the three groups among the patients who received greater than 10 units of PRBC; Test type: Superiority or Other; p = 0.34, test for proportions — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Between May 2006 and August 2009, which was 3 years and 3 months
Description: Serial blood sodium levels were drawn to monitor the effects of the hypertonic saline solutions; Serial head CT's were done to monitor for intracranial hemorrhage
Arm/Group | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline
Serious Adverse Events (participants affected / at risk) | 21/220 | 25/256 | 21/376
Other Adverse Events (participants affected / at risk) | 1/220 | 1/256 | 1/376
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) (N=220) | 7.5% Hypertonic Saline (HS) (N=256) | 0.9% Normal Saline (N=376)
Hypernatremia that required therapeutic intervention (Blood and lymphatic system disorders) | 2 (2) | 5 (5) | 5 (5) — Serum sodium>160 mEq/L requiring therapeutic intervention
Increased intracranial hemorrrhage (Nervous system disorders) | 12 (12) | 14 (14) | 15 (15) — Evidence observed on serial head CT scanning
Hypernatremia that did not required therapeutic intervention (Blood and lymphatic system disorders) | 7 (7) | 6 (6) | 1 (1) — Serum sodium>160 mEq/L that did not require therapeutic intervention
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 7.5% Hypertonic Saline/6% Dextran-70 (HSD) (N=220) | 7.5% Hypertonic Saline (HS) (N=256) | 0.9% Normal Saline (N=376)
Pain, rash, hypotension secondary to a transfusion reaction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — 200 cc red blood cells typed for another patient and not felt to be related to study intervention
Complete placental abruption leading to fetal demise (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) — Protocol violation: enrolled obviously pregnant woman, 6 months gestation
Seizure activity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Observed in prehospital setting during 7.5% hypertonic saline/6% dextran-70 (HSD) fluid administration

LIMITATIONS AND CAVEATS:
The trial was stopped early for futility in the presence of a potential safety concern regarding increased mortality among patients receiving hypertonic solutions and no blood transfusions. This was no longer evident 6 hr after hospital admission.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No